CLINICAL TRIAL: NCT00729794
Title: Vasopressin, Epinephrine, and Corticosteroids for Inhospital Cardiac Arrest: A Multicenter Randomized Controlled Trial
Brief Title: Vasopressin, Epinephrine, and Steroids for Cardiac Arrest
Acronym: VSE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Athens (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Spyros D. Mentzelopoulos, Assistant Professor in Intensive Care Medicine, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VSE-226-2008
Record Dates: First submitted 2008-07-31; First posted 2008-08-08 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Cardiac Arrest
Keywords: Vasopressin; Epinephrine; Adrenal Cortex Hormones; Heart Arrest
MeSH Terms: conditions — Heart Arrest; Diabetes Insipidus | interventions — Vasopressins; Epinephrine; Methylprednisolone; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Experimental): Patients with refractory, inhospital cardiac arrest, i.e., with asystole, pulseless electrical activity, or ventricular fibrillation/pulseless ventricular tachycardia not responsive to two attempts at defibrillation.
  Interventions: Drug: Vasopressin, Epinephrine, Methylprednisolone, Hydrocortisone
- Control Group (Placebo Comparator): Patients with refractory, inhospital cardiac arrest, i.e., with asystole, pulseless electrical activity, or ventricular fibrillation/pulseless ventricular tachycardia not responsive to two attempts at defibrillation.
  Interventions: Drug: Standard CPR Protocol with Epinephrine and two Placebos

INTERVENTIONS:
Drug: Vasopressin, Epinephrine, Methylprednisolone, Hydrocortisone — Combination Treatment
  Administration of vasopressin, epinephrine, and methylprednisolone during CPR, and of stress dose hydrocortisone after CPR
  Arms: Study Group
Drug: Standard CPR Protocol with Epinephrine and two Placebos — Patients receive advanced life support according to the Guidelines for Resuscitation 2005
  Arms: Control Group

SUMMARY:
The simultaneous activation of adrenergic and vasopressin receptors, in conjunction with a potential steroid-mediated enhancement of the vascular reactivity to epinephrine may have beneficial effects in patients with cardiac arrest. This hypothesis is supported by the single-center results of NCT 00411879. The investigators intend to either refute or provide definitive evidence supporting this hypothesis (and its generalizability) by conducting the present multicenter, randomized, controlled clinical trial of in hospital cardiac arrest.

DETAILED DESCRIPTION:
Background and Rationale Inhospital cardiac arrest still constitutes an important clinical problem with survival to discharge ranging within 0-42% (most common range = 15-20%) (1). Survival after witnessed, pulseless ventricular fibrillation/tachycardia (VF/VT) that is responsive to one or two direct current countershock(s) may exceed 30%. However, survival after inhospital asystole, pulseless electrical activity, or refractory VF/VT (defined as not responsive to two countershocks) may be substantially lower (i.e., 5-10%) (2). As in nonsurvivors, both endogenous vasopressin and adrenocorticotrophin are reduced compared to survivors (3,4), the investigators hypothesize that the addition of exogenous vasopressin during cardiopulmonary resuscitation (CPR) (5) and of steroids during and after CPR may increase the rates of return of spontaneous circulation (ROSC) and improve post-arrest survival. This hypothesis is supported by the single-center results of NCT 00411879. Thus, the investigators intend to either refute or provide definitive evidence supporting this hypothesis (and its generalizability) by conducting the present multicenter, randomized, controlled clinical trial of inhospital cardiac arrest.

Methods Adult in-patients with cardiac arrest not responsive to two direct current countershocks (when applicable), or asystole, or pulseless electrical activity are randomized to receive either arginine vasopressin (20 IU/CPR cycle for the first 5 CPR-cycles in non-VF/VT and from the second to sixth CPR-cycle in VF/VT) plus epinephrine (1 mg/CPR-cycle) plus methylprednisolone (single dose = 40 mg during the first and second CPR-cycle in non-VF/VT and VF/VT, respectively) or normal saline-placebo plus epinephrine (1 mg/CPR-cycle) plus normal saline-placebo during the first 5 or second to sixth CPR-cycles. Further CPR-vasopressor treatment includes epinephrine (1 mg/CPR-cycle) for both groups. Apart from the initial, combined drug administration in the study group, CPR is conducted in full concordance with the 2005 Guidelines for Advanced Life Support (5). Following ROSC and in the presence of postresuscitation shock (defined as inability to maintain mean arterial pressure > 70 mm Hg without using exogenous catecholamines at infusion rates conferring vasopressor and/or inotropic activity), study group patients receive stress-dose hydrocortisone (300 mg/day for a maximum of 7 days and then gradual taper), whereas controls receive saline placebo. Patients with pre-arrest history and clinical features, and/or electrocardiographic, biochemical, and echocardiographic evidence of acute myocardial infarction receive the stress-dose hydrocortisone (study-group) or the saline-placebo (control-group) for a maximum of 3 days, followed by gradual taper.1 This time-limit has been chosen to prevent any potential retardation of infarct healing by glucocorticoid treatment (6).

Following ROSC, control group patients may receive stress dose steroid treatment if prescribed by the attending physician for indications such as septic shock or known adrenocortical insufficiency. This holds also for study group patients during the follow-up period. Any steroid prescription by attending physicians cancels any concomitant investigational interventions regarding steroid supplementation and results in patient exclusion, unless the prescribed corticosteroid regimen is in full concordance with the above-described, protocolized one.

The investigators involved in CPR drug administration are blinded to the use (or no-use) of vasopressin and methylprednisolone, and do not coordinate the CPR procedures. For the study group, steroid treatment is determined by the hospital pharmacies, which are also aware of the computer-based patient randomization and encoding, and prepare the study drugs for CPR.

Patient follow-up and data recording is conducted by associates who are unaware of CPR drug regimens. Daily follow-up to day 60 post-arrest includes physiological variables, medication and other treatment interventions, results of laboratory and diagnostic studies (including serum interleukins for days 1-10), and determination of the sequential organ dysfunction assessment (SOFA) score. For the first 10 days post-randomization, monitored/recorded physiological variables include hemodynamics (arterial and central venous pressure, and heart rate), gas exchange and respiratory mechanics, body temperature, urinary output and fluid balance. Patient neurological status will be assessed with the Glasgow Coma Score. Additional follow-up data will include hospital/intensive care unit (ICU)-related morbidity, length of ICU/hospital stay, and cerebral performance/residual disabilities (7) at hospital discharge.

As in previous cardiac arrest trials, the requirement of informed consent for the drug combination during CPR has been waived. However, informed consent is actually requested for corticosteroid treatment of postresuscitation shock. Furthermore, the patients' families are always informed about the trial after the resuscitation procedures. Any next-of-kin objection regarding the trial will result in patient exclusion.

Randomization Technique Randomization will be conducted in blocks of four with the use of the Research Randomizer (www.randomizer.org).

Pre-specified subgroup analyses included the effect of study center, and data from patient subgroups defined according to the need for >5mg or =<5 mg of epinephrine during CPR.

Post hoc analyses included within-group control group comparisons according to the actual use or no use of stress dose hydrocortisone (300 mg /day for a maximum of 7 days followed by gradual taper) by attending physicians. Also, patients without "crossover" of the control group were compared to patients of the VSE group. Lastly, following a relative suggestion by the Data Monitoring Committee, we attempted to determine the 1 year survival with good neurological recovery; for this purpose, survivors of both groups (and/or their families) were contacted / interviewed through telephone communication; this was followed by in-person interview/examination of the survivors.

After completion of three years from the last patient data collection on the primary outcomes, the study data will be maintained in de-identified electronic form.

In concordance with a suggestion of a recent Editorial (Intensive Care Med (2014) 40:743-745), the Original and (its minor revision to) the Final Form of the Study Protocol detailing the Pre-specified Study Planning (which explains the reason for any prior changes in the current registration data) can be found at the bottom of the following webpage: http://www.evaggelismos-hosp.gr/index.php/istoriko-eepne

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with refractory inhospital cardiac arrest, defined as epinephrine requirement for ventricular fibrillation/tachycardia or asystole/pulseless electrical activity according to guidelines for resuscitation 2005 (5).

Exclusion Criteria:

* Age < 18 years
* Terminal illness or do-not resuscitate status
* Cardiac arrest due to exsanguination
* Cardiac arrest before hospital admission
* Pre-arrest treatment with intravenous corticosteroids
* Previous enrollment in or exclusion from the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Return of Spontaneous Circulation for at least 15 min and Survival to Hospital Discharge with or without neurological recovery | 60 days

SECONDARY OUTCOMES:
Arterial pressure and gas exchange during CPR and at 15-20 min following return of spontaneous circulation; hemodynamic status during days 1 to 10 post-randomization | 30 min to 10 days
The number of organ failure-free days during follow-up | 60 days
Complications related to the use of steroids | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Spyros D Mentzelopoulos, MD, PhD, Principal Investigator — University of Athens Medical School, Athens, Greece; Spyros G Zakynthinos, MD, PhD, Study Director — University of Athens Medical School, Athens, Greece; Charis Roussos, MD, PhD, Study Chair — University of Athens Medical School, Athens, Greece
Locations (3):
- Greece (3):
  - Evaggelismos General Hospital, Athens, Attica
  - 401 General Military Hospital of Athens, Athens, Attica
  - University General Hospital of Larissa, Larissa, Thessaly

REFERENCES:
- [Background] Sandroni C, Nolan J, Cavallaro F, Antonelli M. In-hospital cardiac arrest: incidence, prognosis and possible measures to improve survival. Intensive Care Med. 2007 Feb;33(2):237-45. doi: 10.1007/s00134-006-0326-z. Epub 2006 Sep 22. PMID 17019558
- [Background] Stiell IG, Hebert PC, Wells GA, Vandemheen KL, Tang AS, Higginson LA, Dreyer JF, Clement C, Battram E, Watpool I, Mason S, Klassen T, Weitzman BN. Vasopressin versus epinephrine for inhospital cardiac arrest: a randomised controlled trial. Lancet. 2001 Jul 14;358(9276):105-9. doi: 10.1016/S0140-6736(01)05328-4. PMID 11463411
- [Background] Adrie C, Laurent I, Monchi M, Cariou A, Dhainaou JF, Spaulding C. Postresuscitation disease after cardiac arrest: a sepsis-like syndrome? Curr Opin Crit Care. 2004 Jun;10(3):208-12. doi: 10.1097/01.ccx.0000126090.06275.fe. PMID 15166838
- [Background] Hekimian G, Baugnon T, Thuong M, Monchi M, Dabbane H, Jaby D, Rhaoui A, Laurent I, Moret G, Fraisse F, Adrie C. Cortisol levels and adrenal reserve after successful cardiac arrest resuscitation. Shock. 2004 Aug;22(2):116-9. doi: 10.1097/01.shk.0000132489.79498.c7. PMID 15257083
- [Background] Nolan JP, Deakin CD, Soar J, Bottiger BW, Smith G; European Resuscitation Council. European Resuscitation Council guidelines for resuscitation 2005. Section 4. Adult advanced life support. Resuscitation. 2005 Dec;67 Suppl 1:S39-86. doi: 10.1016/j.resuscitation.2005.10.009. No abstract available. PMID 16321716
- [Background] Shizukuda Y, Miura T, Ishimoto R, Itoya M, Iimura O. Effect of prednisolone on myocardial infarct healing: characteristics and comparison with indomethacin. Can J Cardiol. 1991 Dec;7(10):447-54. PMID 1768984
- [Background] A randomized clinical trial of calcium entry blocker administration to comatose survivors of cardiac arrest. Design, methods, and patient characteristics. The Brain Resuscitation Clinical Trial II Study Group. Control Clin Trials. 1991 Aug;12(4):525-45. doi: 10.1016/0197-2456(91)90011-a. PMID 1657528
- [Derived] Holmberg MJ, Granfeldt A, Mentzelopoulos SD, Andersen LW. Vasopressin and glucocorticoids for in-hospital cardiac arrest: A systematic review and meta-analysis of individual participant data. Resuscitation. 2022 Feb;171:48-56. doi: 10.1016/j.resuscitation.2021.12.030. Epub 2022 Jan 3. PMID 34990764
- [Derived] Mentzelopoulos SD, Malachias S, Chamos C, Konstantopoulos D, Ntaidou T, Papastylianou A, Kolliantzaki I, Theodoridi M, Ischaki H, Makris D, Zakynthinos E, Zintzaras E, Sourlas S, Aloizos S, Zakynthinos SG. Vasopressin, steroids, and epinephrine and neurologically favorable survival after in-hospital cardiac arrest: a randomized clinical trial. JAMA. 2013 Jul 17;310(3):270-9. doi: 10.1001/jama.2013.7832. PMID 23860985